CLINICAL TRIAL: NCT03164512
Title: The Pharmacokinetics and Pharmacodynamics of Oral and Vaporized Cannabidiol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00128331
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Cannabidiol Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: placebo controlled, double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo oral and vapor
  Interventions: Drug: Placebo
- Vaporized High Cannabidiol Cannabis (Experimental): Cannabis containing approximately 100mg cannabidiol and 5mg delta-9-THC
  Interventions: Drug: Oral or vaporized cannabidiol
- Vaporized Cannabidiol (Experimental): 100mg cannabidiol in vapor
  Interventions: Drug: Oral or vaporized cannabidiol
- Oral Cannabidiol (Experimental): 100mg oral cannabidiol
  Interventions: Drug: Oral or vaporized cannabidiol

INTERVENTIONS:
Drug: Oral or vaporized cannabidiol — Acute drug exposure
  Arms: Oral Cannabidiol; Vaporized Cannabidiol; Vaporized High Cannabidiol Cannabis
Drug: Placebo — Placebo capsule/vapor
  Arms: Placebo

SUMMARY:
This study will evaluate the pharmacokinetics and pharmacodynamics of cannabidiol administered via inhalation and oral ingestion.

DETAILED DESCRIPTION:
The proposed study will be conducted at the Johns Hopkins Behavioral Pharmacology Research Unit (BPRU) and the Johns Hopkins Bayview Clinical Research Unit (CRU). Participants will complete 4 acute drug administration periods, each consisting of a single drug exposure followed by a 5-day observation period (3-days (58-hours) inpatient and 2-days outpatient). Biological specimens will be obtained to characterize the pharmacokinetics of THC, CBD, and their metabolites in whole blood, oral fluid, urine, and hair during this period. Each participant will receive all 4 dose conditions in a counterbalanced order using a placebo controlled within-subject crossover design. The 4 drug conditions are as follows:

* Condition 1: Inhalation of cannabis vapor containing approximately a 20:1 ratio of CBD:THC and will be measured to deliver a target dose of 100mg CBD and 5mg THC.
* Condition 2: Inhalation of 100mg CBD vapor.
* Condition 3: Ingestion of 100mg CBD.
* Condition 4: Placebo

Drug administration will be double blind and double dummy; both inhalation and oral ingestion of study drugs will occur during all 4 sessions. The order of drug administration will be counterbalanced across participants.

Research volunteers will be recruited until up to 18 participants have completed each of the four study sessions (received Conditions 1-4). Immediately before (baseline) and following each exposure, a battery of assessments including biological fluid collection and testing, subjective questionnaire administration, and performance testing will be conducted for all study participants. Post-exposure testing will be conducted in two phases: a 3-day (58 hour) residential stay, and a 2-day outpatient period, for a total of 5 days. Participants who drop out of the study prior to completion of all 4 drug conditions will be considered "incomplete" and replaced. Approximately one week (minimum of 6 days) will separate the administration of each dose.

The target demographic for study participation are healthy adults who: 1) have a history of intentionally inhaling cannabis/CBD, 2) have not used cannabis in the past month (desire is to have participants free of cannabinoids in biological matrices at the time of initial drug administration), and 3) who are not currently dependent on or seeking treatment for use of cannabis or other psychoactive drugs.

Study outcome variables include quantitative levels of CBD and its primary metabolites, THC and its primary metabolites, results of drug testing procedures conducted in accordance with current federal Mandatory Guidelines for workplace drug testing, subjective drug effect ratings, and performance on behavioral assessments. Biological specimens will be analyzed by an independent laboratory with validated analytical procedures that are specific and accurate for measurement of marijuana constituents and related metabolites. Subjective, cardiovascular and behavioral outcomes will be assessed using multiple regression analyses appropriate for repeated measures testing based on the final characteristics of the data set (e.g. normal distribution, skewness, kurtosis), and correlated with biomarker results of interest.

ELIGIBILITY:
Inclusion Criteria

1. Have provided written informed consent
2. Be between the ages of 18 and 45
3. Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
4. Test negative for recent cannabis use in urine at the screening visit (confirmed by GC/MS laboratory test) and again upon admission for each experimental session
5. Test negative for other drugs of abuse, including alcohol at the screening visit and upon arrival for each experimental session
6. Demonstrate ability to expectorate 3-5 mL of "native" oral fluid over a 5-minute period
7. Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission.
8. Have a body mass index (BMI) in the range of 19 to 36 kg/m2
9. Have head hair that is at least 4 cm (approximately one and a half inches) in length on the back of the head.
10. Blood pressure at Screening Visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
11. Have no allergies to any of the ingredients used to prepare cannabis brownies (chocolate, eggs, wheat, etc.).
12. Report prior experience inhaling cannabis (either via smoking or vaporization).

Exclusion Criteria

1. Non-medical use of psychoactive drugs other than, nicotine, alcohol, or caffeine in the month prior to the Screening Visit;
2. History of or current evidence of significant medical or psychiatric illness judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures.
3. Use of an OTC, systemic or topical drug(s), herbal supplement(s), or vitamin(s) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
4. Use of a prescription medication (with the exception of birth control prescriptions) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
5. Use of hemp seeds or hemp oil in any form in the past 3 months.
6. Use of dronabinol (Marinol) within the past 6 months.
7. History of xerostomia (dry mouth), or the presence of mucositis, gum infection or bleeding, or other significant oral cavity disease or disorder that in the investigator's opinion may affect the collection of oral fluid samples.
8. History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
THC-COOH in Urine | Hour 4
  THC-COOH in Urine

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual biological testing data will be published. Requests for additional data can be submitted to Dr. Vandrey via e-mail.
Supporting Information: CSR
Time Frame: Will be available indefinitely after publication of study findings
Access Criteria: Request to the study PI